CLINICAL TRIAL: NCT02517671
Title: Impact of Enhanced External Counterpulsation (EECP) on VO2 MAX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI failed to file continuation report.
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG20140034H
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Disease; Pulmonary Disease
Keywords: Fitness; Run time; VO2max; VEGF; Central blood pressure; Augmentation Index; Pulse wave analysis
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EECP Treatment (Other): 35 one hour (1hr) sessions of Enhanced External Counterpulsation (EECP).
  Interventions: Device: Enhanced External Counterpulsation (EECP)

INTERVENTIONS:
Device: Enhanced External Counterpulsation (EECP) — EECP is a non-invasive therapy that has been approved by the United States Food and Drug Administration (FDA) for the management of refractory angina and heart failure. This study is using the device to potentially improve 1.5 mile run times and VO2max in healthy volunteers.

SUMMARY:
The purpose of this study is to assess the effects of 35 EECP sessions on cardiopulmonary training performance in healthy volunteers. Data from this study will be used to generate sample size and power calculations for feasibility of future EECP studies. The results of this study could provide evidence that can help active duty and Department of Defense beneficiaries optimize physical conditioning, endurance and overall health.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effects of 35 EECP sessions on cardiopulmonary training performance in healthy volunteers. Prior published and anecdotal evidence suggests that EECP should improve athletic performance. Data from this study will be used to generate sample size and power calculations for feasibility of future EECP studies. The results of this study could provide evidence that can help active duty and Department of Defense beneficiaries optimize physical conditioning, endurance and overall health. It could help active duty members maximize their physical training potential enabling them to better prepare for missions down range. Additionally, physiologic cardiopulmonary improvements may have the potential to decrease the conditioning time required for injured, post-operative and post-partum active duty members to return to duty.

ELIGIBILITY:
Inclusion Criteria:

* Healthy active-duty military personnel or DoD beneficiaries

  * Medically cleared for the 1.5 mile run test [subjects will be medically cleared via PI's discretion or physician consultation letter]
* 18 years or older [no age cutoff is needed, subjects will be medically cleared via PI's discretion or physician consultation letter]
* Scoring below 55 out of 60 points on a 1.5 mile run portion of test using current AFI fitness standards [adjusted for age and gender]
* Maintaining a steady work-out routine and agreeing to adhere to it for the duration of the study. The workouts cannot vary by greater than 50% week to week (e.g. a subject that works out 3 hours on week 1, can only work out between 1.5 to 4.5 hours on week 2).
* Dermatological conditions not impacted by the EECP procedure will be allowed to enroll (e.g. eczema).

Exclusion Criteria:

* Pregnancy or anticipated pregnancy
* Exemption from PT (run portion of physical fitness test)
* VO2MAX greater than 55 mL/kg/min [determined from baseline CPX]
* Scheduled permanent change in station within 3 months
* Any significant co-morbid health conditions medically classifying the subject as not healthy [at PI's discretion], including but not limited to the following.

  * Previous myocardial infarction, hernias, aneurysms, retinal detachments (unless fixed by laser surgery), macular edema, chest pain, ocular bleeding or seizures
  * Risk of pulmonary edema
  * Diagnosed with diabetes, heart failure, atrial fibrillation or epilepsy
  * Coagulopathy with an INR of prothrombin time > 2.5
  * Valvular heart disease
  * Blood pressure >140/100 mmHg or <90/60 mmHg upon clinic visit
  * Subjects with heart rates >120 bpm upon clinic visit
  * Subjects with implantable cardioverter-defibrillator or pacemaker
  * History of deep vein thrombosis
  * History of pulmonary embolism
  * Family history of individuals with multiple pulmonary embolisms or young onset pulmonary embolism (< 65 years old)
  * Bleeding diathesis
  * Presence of abdominal surgery within the past 6 months in EMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10-07 (Estimated); Study Completion 2017-10-07 (Actual)

PRIMARY OUTCOMES:
VO2 MAX | 7 weeks
  The primary endpoint will be the change from baseline in VO2 MAX over the 7-week EECP treatment period.

SECONDARY OUTCOMES:
1.5 run run | 7 weeks
  The secondary endpoint will be the change in 1.5 mile run time pre/post a 7-week course of EECP therapy.

OTHER OUTCOMES:
Exploratory endpoints peripheral blood pressures | 7 weeks
  Assessment of peripheral blood pressures levels.
Exploratory endpoints Central Blood Pressure | 7 weeks
  Assessment of Central Blood Pressure levels
Exploratory endpoints Augmentation index | 7 weeks
  Assessment of Augmentation index
Exploratory endpoints VEGF | 7 weeks
  Assessment of VEGF

CONTACTS AND LOCATIONS:
Overall Officials: Sokunthea Peou, Pharmacist, Principal Investigator — David Grant Medical Center
Locations (1):
- David Grant AF Medical Center, Travis Air Force Base, California, United States